CLINICAL TRIAL: NCT00424593
Title: Effect of Duloxetine 60 mg to 120 mg Once Daily in Patients With Chronic Low Back Pain
Brief Title: Duloxetine Versus Placebo in Chronic Low Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10544; F1J-MC-HMEN
Record Dates: First submitted 2007-01-17; First posted 2007-01-19 (Estimated); Results first posted 2009-11-18 (Estimated); Last update posted 2009-11-20 (Estimated); Status verified 2009-11

CONDITIONS: Back Pain Without Radiation
MeSH Terms: conditions — Back Pain | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Duloxetine (Experimental): 30 mg, every day (QD), by mouth (PO) for 1 week followed by 60 mg, QD, PO, 6 weeks then 60 mg (responders) or 120 mg (non-responders), QD, PO, 6 weeks during the placebo-controlled phase, then 60 mg or 120 mg, QD, PO, 41 weeks during the extension phase
  Interventions: Drug: Duloxetine
- Placebo (Placebo Comparator): every day (QD), by mouth (PO), 13 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Duloxetine — 30 mg, every day (QD), by mouth (PO) for 1 week followed by 60 mg, QD, PO, 6 weeks then 60 mg (responders) or 120 mg (non-responders), QD, PO, 6 weeks during the placebo-controlled phase, then 60 mg or 120 mg, QD, PO, 41 weeks during the extension phase
  Other Names: LY248686; Cymbalta
  Arms: Duloxetine
Drug: Placebo — every day (QD), by mouth (PO), 13 weeks
  Arms: Placebo

SUMMARY:
The primary purpose of your participation in this study is to help answer the following research question, and not to provide you treatment for your condition.

Whether duloxetine once daily can help patients with Chronic Low Back Pain.

Patients who do not have their pain reduced by at least 30% by week 7 will be given 120 mg dose for the duration of the study. After the 13 week double blind period, patients randomized to placebo will switch to duloxetine 60 mg or 120 mg in the 41-week extension period.

ELIGIBILITY:
Inclusion Criteria:

* Male/Female outpatients 18 years of age with chronic low back pain
* Females of child bearing potential must test negative on a pregnancy test at visit 1.

Exclusion Criteria:

* Have a serious or unstable diseases of the heart or blood vessels, liver, kidney, lungs, or blood-related illness
* Problems with decreased blood flow to arms and legs (peripheral vascular disease), or other medical conditions
* Psychiatric conditions that, in the opinion of the investigator, would affect your participation or be likely to lead to hospitalization during the course of the study
* Have acute liver injury (such as hepatitis) or severe cirrhosis
* Have had previous exposure to duloxetine
* Have a body mass index (BMI) over 40
* Have a major depressive disorder
* Require daily narcotics
* Have suicidal risk
* Have a presence of any factors/conditions, medical or other, that in the judgment of the investigator may interfere with performance of study outcome measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2007-01; Primary Completion 2007-12 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (16):
- Brazil (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your p, Curitiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your p, São Paulo
- France (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your p, Amiens
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your p, Marseille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your p, Paris
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your p, Saint-Affrique
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your p, Saint-Etienne
- Germany (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your p, Ellwangen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your p, Gräfelfing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your p, Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your p, Wiesbaden
- Mexico (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your p, Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your p, Monterrey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your p, San Pedro Garza García
- Netherlands (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your p, Amsterdam
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your p, Rotterdam

REFERENCES:
- [Derived] Williamson OD, Schroer M, Ruff DD, Ahl J, Margherita A, Sagman D, Wohlreich MM. Onset of response with duloxetine treatment in patients with osteoarthritis knee pain and chronic low back pain: a post hoc analysis of placebo-controlled trials. Clin Ther. 2014 Apr 1;36(4):544-51. doi: 10.1016/j.clinthera.2014.02.009. Epub 2014 Mar 17. PMID 24650448
- [Derived] Skljarevski V, Zhang S, Chappell AS, Walker DJ, Murray I, Backonja M. Maintenance of effect of duloxetine in patients with chronic low back pain: a 41-week uncontrolled, dose-blinded study. Pain Med. 2010 May;11(5):648-57. doi: 10.1111/j.1526-4637.2010.00836.x. Epub 2010 Apr 13. PMID 20546509
- [Derived] Skljarevski V, Desaiah D, Liu-Seifert H, Zhang Q, Chappell AS, Detke MJ, Iyengar S, Atkinson JH, Backonja M. Efficacy and safety of duloxetine in patients with chronic low back pain. Spine (Phila Pa 1976). 2010 Jun 1;35(13):E578-85. doi: 10.1097/BRS.0b013e3181d3cef6. PMID 20461028
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Period: Acute Double-Blind Period
Arm/Group | Duloxetine | Placebo
Started | 115 | 121
Completed | 84 | 98
Not Completed | 31 | 23
Not completed — Adverse Event | 16 | 7
Not completed — Withdrawal by Subject | 11 | 10
Not completed — Protocol Violation | 2 | 2
Not completed — Physician Decision | 1 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Lack of Efficacy | 0 | 1
Period: Dose-Blind Extension Period
Arm/Group | Duloxetine | Placebo
Started | 181 (83 duloxetine patients from the acute phase entered the dose-blind period.) | 0 (98 placebo patients from acute phase entered dose-blind period and received duloxetine.)
Completed | 117 | 0
Not Completed | 64 | 0
Not completed — Withdrawal by Subject | 19 | 0
Not completed — Adverse Event | 18 | 0
Not completed — Lack of Efficacy | 9 | 0
Not completed — Protocol Violation | 9 | 0
Not completed — Lost to Follow-up | 6 | 0
Not completed — Physician Decision | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Duloxetine | Placebo | Total
Number analyzed (Participants) | 115 | 121 | 236
Age Continuous [Mean (Standard Deviation); unit: years] | 51.81 (14.92) | 51.15 (13.46) | 51.47 (14.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 73 | 144
  Male | 44 | 48 | 92
Region of Enrollment [Number; unit: participants]
  France | 11 | 12 | 23
  Mexico | 23 | 20 | 43
  Brazil | 25 | 29 | 54
  Netherlands | 19 | 25 | 44
  Germany | 37 | 35 | 72
Race/Ethnicity [Number; unit: participants]
  African | 6 | 6 | 12
  Caucasian | 85 | 91 | 176
  East Asian | 0 | 2 | 2
  Hispanic | 23 | 21 | 44
  Native American | 1 | 1 | 2
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per square meter (kg/m^2)] — Body mass index is an estimate of body fat based on body weight divided by height squared.
  kilograms per square meter (kg/m^2) | 27.63 (4.42) | 27.03 (3.81) | 27.33 (4.12)
Brief Pain Inventory (BPI) Average Pain Score [Mean (Standard Deviation); unit: units on a scale] — A self-reported scale that measures the severity of pain based on the average pain over the past 24-hours. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine).
  units on a scale | 5.91 (1.59) | 5.96 (1.66) | 5.94 (1.62)
Duration of Chronic Lower Back Pain Since Onset [Mean (Standard Deviation); unit: years] | 8.79 (8.75) | 9.54 (8.60) | 9.18 (8.66)
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 165.92 (10.39) | 167.40 (11.34) | 166.68 (10.89)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 76.24 (14.71) | 75.89 (13.94) | 76.06 (14.29)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 13 in Brief Pain Inventory (BPI), 24-hour Average Pain Scores
Description: A self-reported scale that measures the severity of pain based on the average pain over the past 24-hours. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine).
Time Frame: Baseline, Week 13
Population: Number of participants with baseline and at least one non-missing post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 109 | 115
units on a scale | -2.32 (0.22) | -1.50 (0.21)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.004, Repeated Measures Analysis — Model included treatment, non-steriodal anti-inflammatory drug (NSAID) use (Yes/No), investigator, visit, treatment-by-visit interaction, baseline pain severity, and baseline-by-visit interaction

2. Secondary Outcome: Patient's Global Impression of Improvement (PGI-I)
Description: A scale that measures the patient's perception of improvement at the time of assessment. The score ranges from 1 (very much better) to 7 (very much worse).
Time Frame: Week 13
Population: Number of participants with at least one non-missing post-baseline value. Last observation carried forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 107 | 115
units on a scale | 2.81 (1.18) | 3.23 (1.26)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.014, ANCOVA

3. Secondary Outcome: Change From Baseline to Week 13 and Week 54 Endpoints in Roland Morris Disability Questionnaire-24 Item (RMDQ-24) Total Score
Description: Roland-Morris questionnaire will be completed by the patient and measures the degree of disability due to back pain. The questionnaire consists of 24 statements and the patient is instructed to put a mark next to each appropriate statement. The number of statements marked will be added up by the clinician and a total score is given. The total score ranges from 0 (no disability) to 24 (severe disability).
Time Frame: Baseline, Week 13, Week 54
Population: Number of participants with a baseline and at least one non-missing post-baseline value. Last observation carried forward.
  Note: Week 54 was the end of the extension phase and all patients received duloxetine - data are reported per the original randomized group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 99 | 105
units on a scale
  13 Week Baseline | 10.39 (4.78) | 10.87 (5.12)
  13 Week Change from Baseline | -3.13 (4.65) | -1.53 (4.85)
  54 Week Baseline (n=59, n=82) | 7.83 (5.75) | 9.59 (6.11)
  54 Week Change from Baseline (n=59, n=82) | -1.14 (3.51) | -2.40 (5.30)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.009, ANCOVA — P-value is for 13 Week Change from Baseline

4. Secondary Outcome: Change From Baseline to Week 13 Endpoint in Weekly Mean of 24-hour Average Pain, Night Pain and Worst Pain by 11-Point Likert Scale
Description: 24-hour average pain severity scores recorded daily on an 11-point Likert scale, an ordinal scale ranging from 0 (no pain) to 10 (worst possible pain). Patients should complete the electronic diary at bedtime. The 11-point Likert scale will also be used for assessment of night pain and worst pain each day, and evaluated as weekly means. Average interference was calculated as the average of non-missing scores of individual interference items.
Time Frame: Baseline, Week 13
Population: Number of randomized participants with a baseline and at least one non-missing post-baseline value. Last observation carried forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 111 | 116
units on a scale
  Average Pain Score Baseline | 5.94 (1.36) | 6.05 (1.33)
  Average Pain Score Change from Baseline | -1.92 (1.91) | -1.16 (1.95)
  Worst Pain Score Baseline | 6.91 (1.24) | 7.02 (1.21)
  Worst Pain Score Change from Baseline | -1.97 (2.01) | -1.31 (1.89)
  Night Pain Score Baseline | 5.46 (1.77) | 5.50 (1.81)
  Night Pain Score Change from Baseline | -1.82 (2.01) | -1.15 (1.94)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.002, ANCOVA — P-value for Average Pain Score Change from Baseline
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.014, ANCOVA — P-value for Worst Pain Score Change from Baseline
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.007, ANCOVA — P-value for Night Pain Score Change from Baseline

5. Secondary Outcome: Change From Baseline to Week 13 and Week 54 Endpoints in Brief Pain Inventory - Severity (BPI-S) and Interference (BPI-I) Scores
Description: BPI-S and BPI-I are self-reported scales measuring severity of pain and interference on function. Severity scores: 0 (no pain) to 10 (severe pain) on each question assessing worst pain, least pain, and average pain in past 24 hours, and pain right now. Interference scores: 0 (does not interfere) to 10 (completely interferes) on each question assessing interference of pain in past 24 hours for general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. Average interference = average of non-missing scores of individual interference items.
Time Frame: Baseline, Week 13, Week 54
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 109 | 115
units on a scale
  Worst Pain Score Week 13 Baseline | 7.43 (1.34) | 7.34 (1.46)
  Worst Pain Score Week 13 Change from Baseline | -2.55 (2.31) | -1.72 (2.25)
  Worst Pain Score Week 54 Baseline (n=80, n=97) | 4.49 (2.14) | 5.67 (2.38)
  Worst Pain Score Week 54 Change from Baseline | -1.31 (2.43) | -1.78 (2.56)
  Least Pain Score Week 13 Baseline | 4.22 (2.33) | 4.22 (2.42)
  Least Pain Score Week 13 Change from Baseline | -1.72 (2.05) | -0.83 (2.16)
  Least Pain Score Week 54 Baseline (n=80, n=97) | 2.36 (1.98) | 3.33 (2.60)
  Least Pain Score Week 54 Change from Baseline | -0.81 (1.67) | -0.93 (2.21)
  Average Pain Score Week 13 Baseline | 5.91 (1.61) | 5.93 (1.67)
  Average Pain Score Week 13 Change from Baseline | -2.08 (2.14) | -1.43 (2.25)
  Average Pain Score Week 54 Baseline (n=80, n=97) | 3.40 (1.87) | 4.45 (2.29)
  Average Pain Score Week 54 Change from Baseline | -1.05 (1.79) | -1.35 (2.24)
  Pain Right Now Score Week 13 Baseline | 5.42 (2.12) | 5.55 (2.05)
  Pain Right Now Score Week 13 Change from Baseline | -2.29 (2.41) | -1.43 (2.53)
  Pain Right Now Score Week 54 Baseline (n=80, n=97) | 2.75 (1.96) | 4.11 (2.58)
  Pain Right Now Score Week 54 Change from Baseline | -0.76 (2.01) | -1.25 (2.48)
  General Activity Week 13 Baseline | 5.07 (2.26) | 5.60 (2.29)
  General Activity Week 13 Change from Baseline | -1.83 (2.57) | -1.51 (2.86)
  General Activity Week 54 Baseline (n=80, n=97) | 3.11 (2.34) | 4.05 (2.78)
  General Activity Week 54 Change from Baseline | -0.86 (2.10) | -1.32 (2.78)
  Mood Week 13 Baseline | 3.89 (2.56) | 4.30 (2.76)
  Mood Week 13 Change from Baseline | -1.70 (2.73) | -1.03 (3.24)
  Mood Week 54 Baseline (n=80, n=97) | 1.89 (2.33) | 3.24 (3.00)
  Mood Week 54 Change from Baseline | -0.44 (2.19) | -0.93 (2.69)
  Walking Ability Week 13 Baseline | 4.49 (2.66) | 4.83 (2.76)
  Walking Ability Week 13 Change from Baseline | -2.01 (2.91) | -1.34 (2.94)
  Walking Ability Week 54 Baseline (n=80, n=97) | 2.49 (2.61) | 3.53 (2.83)
  Walking Ability Week 54 Change from Baseline | -0.51 (2.14) | -1.27 (2.62)
  Normal Work Week 13 Baseline | 5.01 (2.39) | 5.39 (2.39)
  Normal Work Week 13 Change from Baseline | -2.10 (2.66) | -1.58 (3.12)
  Normal Work Week 54 Baseline (n=80, n=97) | 2.85 (2.49) | 3.81 (2.72)
  Normal Work Week 54 Change from Baseline | -0.71 (2.18) | -1.09 (2.32)
  Relations With People Week 13 Baseline | 2.75 (2.57) | 3.39 (2.91)
  Relations With People Week 13 Change from Baseline | -1.28 (2.76) | -0.92 (3.37)
  Relations With People Week 54 Baseline (n=80,n=97) | 1.48 (1.99) | 2.53 (2.69)
  Relations With People Week 54 Change from Baseline | -0.51 (1.44) | -0.77 (2.57)
  Sleep Week 13 Baseline | 4.12 (2.81) | 4.59 (2.64)
  Sleep Week 13 Change from Baseline | -1.66 (3.19) | -1.30 (3.01)
  Sleep Week 54 Baseline (n=80, n=97) | 2.38 (2.38) | 3.40 (2.81)
  Sleep Week 54 Change from Baseline | -1.13 (2.31) | -1.08 (2.38)
  Enjoyment of Life Week 13 Baseline | 3.57 (2.84) | 3.41 (2.74)
  Enjoyment of Life Week 13 Change from Baseline | -1.72 (2.82) | -0.81 (2.96)
  Enjoyment of Life Week 54 Baseline (n=80, n=97) | 1.61 (2.22) | 2.61 (2.91)
  Enjoyment of Life Week 54 Change from Baseline | -0.70 (2.03) | -0.93 (2.33)
  Average Interference Week 13 Baseline | 4.13 (1.92) | 4.50 (2.08)
  Average Interference Week 13 Change from Baseline | -1.76 (2.04) | -1.21 (2.39)
  Average Interference Week 54 Baseline (n=80, n=97) | 2.26 (1.86) | 3.31 (2.34)
  Average Interference Week 54 Change from Baseline | -0.69 (1.39) | -1.06 (1.96)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.011, ANCOVA — P-value for Worst Pain Score Week 13 Change from Baseline
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.001, ANCOVA — P-value for Least Pain Score Week 13 Change from Baseline
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.019, ANCOVA — P-value for Average Pain Score Week 13 Change from Baseline
Statistical Analysis 4: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.002, ANCOVA — P-value for Pain Right Now Score Week 13 Change from Baseline
Statistical Analysis 5: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.068, ANCOVA — P-value for General Activity Week 13 Change from Baseline
Statistical Analysis 6: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.009, ANCOVA — P-value for Mood Week 13 Change from Baseline
Statistical Analysis 7: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.006, ANCOVA — P-value for Walking Ability Week 13 Change from Baseline
Statistical Analysis 8: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.024, ANCOVA — P-value for Normal Work Week 13 Change from Baseline
Statistical Analysis 9: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.005, ANCOVA — P-value for Relations With People Week 13 Change from Baseline
Statistical Analysis 10: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.051, ANCOVA — P-value for Sleep Week 13 Change from Baseline
Statistical Analysis 11: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.013, ANCOVA — P-value for Enjoyment of Life Week 13 Change from Baseline
Statistical Analysis 12: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.005, ANCOVA — P-value for Average Interference Week 13 Change from Baseline

6. Secondary Outcome: Change From Baseline to Week 13 and Week 54 Endpoints in Clinical Global Impression of Severity (CGI-Severity)
Description: Measures severity of illness at the time of assessment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill patients).
Time Frame: Baseline, Week 13, Week 54
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 110 | 117
units on a scale
  Week 13 Baseline | 3.23 (1.51) | 3.27 (1.45)
  Week 13 Change from Baseline | -0.94 (1.29) | -0.74 (1.22)
  Week 54 Baseline (n=81, n=97) | 2.21 (1.15) | 2.60 (1.27)
  Week 54 Change from Baseline (n=81, n=97) | -0.23 (0.84) | -0.52 (1.08)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.092, ANCOVA — P-value for Week 13 Change from Baseline

7. Secondary Outcome: Number of Participants Who Responded to Treatment at Week 13 Endpoint Based on 30% Score Reduction Criteria
Description: Response to treatment was defined as at least a 30% reduction of weekly mean score in in Brief Pain Inventory (BPI) Average Pain severity ratings from baseline to endpoint. The number of participants who met this criteria are presented.
Time Frame: Week 13
Population: Number of randomized participants with non-missing response values.
Measure: Number; unit: participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 109 | 115
participants | 58 | 46
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.060, Fisher Exact

8. Secondary Outcome: Number of Participants Who Responded to Treatment at Week 13 Endpoint Based on 50% Score Reduction Criteria
Description: Response to treatment was defined as at least a 50% reduction of weekly mean score in in Brief Pain Inventory (BPI) Average Pain severity ratings from baseline to endpoint. The number of participants who met this criteria are presented.
Time Frame: Week 13
Population: Number of randomized participants with non-missing response values.
Measure: Number; unit: participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 109 | 115
participants | 42 | 31
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.087, Fisher Exact

9. Secondary Outcome: Change From Baseline to Week 13 and Week 54 Endpoints in Athens Insomnia Scale
Description: Estimates sleep difficulty. Consists of 8 items rated on a 4-point scale of 0 (no problem at all) to 3 (very serious problem). Total score of the 8-item version ranges from 0-24.
Time Frame: Baseline, Week 13, Week 54
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 104 | 106
units on a scale
  Week 13 Baseline | 8.03 (4.63) | 8.29 (5.26)
  Week 13 Change from Baseline | -2.01 (4.62) | -1.50 (5.05)
  Week 54 Baseline (n=71, n=86) | 5.42 (4.44) | 6.70 (5.05)
  Week 54 Change from Baseline (n=71, n=86) | -0.37 (4.32) | -1.05 (4.49)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.329, ANCOVA — P-value for Week 13 Change from Baseline

10. Secondary Outcome: Change From Baseline to Week 13 Endpoint in 36-Item Short-Form Health Survey (SF-36)
Description: The SF-36 Health Status Survey is a generic, health-related scale assessing subjects' quality of life on 8 domains: physical functioning, social functioning, bodily pain, vitality, mental health, role-physical, role-emotional and general health and 2 summary scores (mental component summary [MCS] and physical component summary [PCS]). MCS and PCS scores=0-100 (higher scores indicate better health status). Domain scores: general health=5-25; physical functioning=10-30; role-physical=4-8; role-emotional=3-6; social functioning=2-10; bodily pain=2-11; vitality=4-24; mental health=5-30.
Time Frame: Baseline, Week 13
Population: Number of participants with a baseline and at least one non-missing post-baseline value. Last observation carried forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 102 | 106
units on a scale
  Mental Component Summary Baseline | 49.69 (9.99) | 49.60 (11.11)
  Mental Component Summary Change from Baseline | 2.05 (9.90) | -0.49 (10.45)
  Physical Component Summary Baseline | 33.39 (7.61) | 32.62 (7.37)
  Physical Component Summary Change from Baseline | 5.69 (9.17) | 4.12 (8.97)
  Bodily Pain Baseline | 5.48 (1.38) | 5.42 (1.39)
  Bodily Pain Change from Baseline | 1.55 (2.04) | 0.95 (1.91)
  General Health Baseline | 16.27 (4.00) | 15.75 (4.03)
  General Health Change from Baseline | 1.73 (3.57) | 0.82 (4.08)
  Mental Health Baseline | 22.06 (4.51) | 21.95 (4.52)
  Mental Health Change from Baseline | 1.19 (4.12) | 0.28 (4.58)
  Physical Functioning Baseline | 19.53 (4.26) | 19.87 (4.31)
  Physical Functioning Change from Baseline | 2.59 (4.51) | 1.61 (4.26)
  Role-Emotional Baseline | 4.57 (1.29) | 4.67 (1.31)
  Role-Emotional Change from Baseline | 0.44 (1.41) | 0.12 (1.37)
  Role-Physical Baseline | 5.24 (1.41) | 5.07 (1.33)
  Role-Physical Change from Baseline | 0.63 (1.75) | 0.48 (1.63)
  Social Functioning Baseline | 7.83 (1.77) | 7.57 (1.98)
  Social Functioning Change from Baseline | 0.51 (1.93) | 0.14 (2.08)
  Vitality Baseline | 15.16 (3.33) | 14.79 (3.69)
  Vitality Change from Baseline | 1.08 (3.93) | 0.21 (4.31)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.051, ANCOVA — P-value for Mental Component Summary Change from Baseline
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.220, ANCOVA — P-value for Physical Component Summary Change from Baseline
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.038, ANCOVA — P-value for Bodily Pain Change from Baseline
Statistical Analysis 4: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.041, ANCOVA — P-value for General Health Change from Baseline
Statistical Analysis 5: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.093, ANCOVA — P-value for Mental Health Change from Baseline
Statistical Analysis 6: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.210, ANCOVA — P-value for Physical Functioning Change from Baseline
Statistical Analysis 7: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.170, ANCOVA — P-value for Role-Emotional Change from Baseline
Statistical Analysis 8: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.306, ANCOVA — P-value for Role-Physical Change from Baseline
Statistical Analysis 9: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.053, ANCOVA — P-value for Social Functioning Change from Baseline
Statistical Analysis 10: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.040, ANCOVA — P-value for Vitality Change from Baseline

11. Secondary Outcome: Change From Baseline to Week 13 Endpoint in EuroQoL Questionnaire - 5 Dimension (EQ-5D)
Description: The EuroQoL Questionnaire - 5 Dimension (EQ-5D) is a generic, multidimensional, health-related, quality-of-life instrument. The profile allows patients to rate their health state in 5 health domains: mobility, self-care, usual activities, pain/discomfort, and mood. A single score between 1 and 3 is generated for each domain. For each patient, the outcome rating on the 5 domains will be mapped to a single index through an algorithm. The index ranges between 0 and 1, with the higher score indicating a better health state perceived by the patient. Scores presented used the UK Based Index Score.
Time Frame: Baseline, Week 13
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 101 | 102
units on a scale
  Baseline | 0.49 (0.31) | 0.49 (0.32)
  Change from Baseline | 0.16 (0.32) | 0.11 (0.30)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.117, ANCOVA — P-value for Change from Baseline

12. Secondary Outcome: Change From Baseline to Week 13 and Week 54 Endpoints in Work Productivity and Activity Impairment Instrument (WPAI) Scores
Description: WPAI: self-administered instrument used to measure effect of general health and symptom severity on work productivity and regular activities and yields 4 types of scores: Absenteeism (work time missed); Presenteeism (impairment at work/reduced on-the-job effectiveness); Work Productivity Loss (overall work impairment/absenteeism plus presenteeism); and Activity Impairment. Higher scores are indicative of greater impairment.
  1. Absenteeism=(Q2/(Q2+Q4))*100
  2. Presenteeism=(Q5/10)*100
  3. Work productivity loss=(Q2/(Q2+Q4)+[(1-Q2/(Q2+Q4))x(Q5/10)])*100
  4. Activity Impairment=(Q6/10)*100
Time Frame: Baseline, Week 13, Week 54
Population: Number of participants currently being paid to work who had a baseline and at least one non-missing post-baseline value. Last observation carried forward.
  Note: Week 54 was the end of the extension phase and all patients received duloxetine - data are reported per the original randomized group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 103 | 105
units on a scale
  Absenteeism Score Week 13 Baseline (n=35, n=32) | 0.17 (0.30) | 0.05 (0.10)
  Absenteeism Score Week 13 Change from Baseline | -0.14 (0.29) | 0.03 (0.20)
  Absenteeism Score Week 54 Baseline (n=24, n=32) | 0.03 (0.10) | 0.02 (0.07)
  Absenteeism Score Week 54 Change from Baseline | 0.01 (0.12) | 0.01 (0.14)
  Presenteeism Score Week 13 Baseline (n=37, n=31) | 0.42 (0.30) | 0.36 (0.19)
  Presenteeism Score Week 13 Change from Baseline | -0.17 (0.32) | -0.06 (0.21)
  Presenteeism Score Week 54 Baseline (n=24, n=34) | 0.19 (0.16) | 0.30 (0.25)
  Presenteeism Score Week 54 Change from Baseline | -0.05 (0.20) | -0.13 (0.17)
  Work Productivity Loss Week 13 Baseline(n=33,n=29) | 0.47 (0.31) | 0.38 (0.18)
  Work Productivity Loss Week 13 Change | -0.19 (0.30) | -0.06 (0.21)
  Work Productivity Loss Week 54 Baseline(n=24,n=32) | 0.21 (0.19) | 0.32 (0.26)
  Work Productivity Loss Week 54 Change | -0.04 (0.22) | -0.13 (0.19)
  Activity Impairment Week 13 Baseline (n=103,n=105) | 0.54 (0.23) | 0.57 (0.22)
  Activity Impairment Week 13 Change from Baseline | -0.20 (0.29) | -0.11 (0.25)
  Activity Impairment Week 54 Baseline (n=70, n=86) | 0.32 (0.24) | 0.45 (0.27)
  Activity Impairment Week 54 Change from Baseline | -0.06 (0.20) | -0.16 (0.22)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.063, ANCOVA — P-value for Absenteeism Week 13 Change from Baseline
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.452, ANCOVA — P-value for Presenteeism Week 13 Change from Baseline
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.736, ANCOVA — P-value for Work Productivity Loss Week 13 Change from Baseline
Statistical Analysis 4: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.002, ANCOVA — P-value for Work Activity Impairment Week 13 Change from Baseline

13. Secondary Outcome: Change From Baseline to Week 13 and Week 54 Endpoints in Beck Depression Inventory (BDI-II) Total Scores
Description: A 21-item, patient-completed questionnaire to assess characteristics of depression. Each of the 21 items corresponding to a symptom of depression is summed to give a single score. There is a four-point scale for each item ranging from 0 to 3. Total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe.
Time Frame: Baseline, Week 13, Week 54
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 109 | 116
units on a scale
  Week 13 Baseline | 6.94 (7.73) | 6.81 (6.77)
  Week 13 Change from Baseline | -0.51 (5.50) | 0.68 (6.81)
  Week 54 Baseline (n=80, n=97) | 5.93 (7.18) | 7.69 (9.01)
  Week 54 Change from Baseline (n=80, n=97) | -0.64 (3.98) | -1.01 (6.59)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.177, ANCOVA — P-value for Week 13 Change from Baseline

14. Secondary Outcome: Change From Baseline to Week 13 Endpoint in Hospital Anxiety and Depression Scale (HADS) Scores
Description: A 14-item questionnaire with 2 subscales: anxiety and depression. Each item is rated on a 4-point scale, giving maximum scores of 21 for anxiety and depression. Scores of 11 or more on either subscale are considered to be a significant 'case' of psychological morbidity, while scores of 8-10 represent 'borderline' and 0-7, 'normal.'
Time Frame: Baseline, Week 13
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 103 | 105
units on a scale
  Anxiety Subscale Baseline (n=102, n=104) | 4.94 (3.76) | 4.41 (3.67)
  Anxiety Subscale Change from Baseline | -0.70 (3.18) | 0.11 (3.34)
  Depression Subscale Baseline (n=103, n=105) | 3.65 (3.22) | 3.87 (3.42)
  Depression Subscale Change from Baseline | -0.27 (2.58) | 0.10 (2.99)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.122, ANCOVA — P-value for Anxiety Subscale Change from Baseline
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.262, ANCOVA — P-value for Depression Subscale Change from Baseline

15. Secondary Outcome: Laboratory Assessments That Were Statistically Significantly Different Between Treatment Groups in Change From Baseline to Week 13 Endpoint: Bicarbonate
Time Frame: Baseline, Week 13
Population: Number of participants with a baseline and at least one non-missing post-baseline value, based on the first values at scheduled visits only. Last observation carried forward.
Measure: Mean (Standard Deviation); unit: millimole per Liter (mmol/L)
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 102 | 110
millimole per Liter (mmol/L)
  Baseline | 24.90 (2.80) | 25.10 (2.94)
  Change from Baseline | 0.57 (2.89) | -0.28 (2.84)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.046, ANOVA — P-value for Change from Baseline; ANOVA based on rank transformation

16. Secondary Outcome: Laboratory Assessments That Were Statistically Significantly Different Between Treatment Groups in Change From Baseline to Week 13 Endpoint: Uric Acid
Time Frame: Baseline, Week 13
Population: Number of participants with a baseline and at least one non-missing post-baseline value, based on first values at scheduled visits only. Last observation carried forward.
Measure: Mean (Standard Deviation); unit: micromole per Liter (μmol/L)
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 104 | 111
micromole per Liter (μmol/L)
  Baseline | 303.23 (79.04) | 298.07 (82.63)
  Change from Baseline | -6.27 (37.81) | 8.68 (43.72)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.008, ANOVA — P-value for Change from Baseline; ANOVA based on rank transformation

17. Secondary Outcome: Change From Baseline to Week 13 and Week 54 Endpoints in Vital Signs: Pulse Rate
Time Frame: Baseline, Week 13, Week 54
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 109 | 115
beats per minute (bpm)
  Week 13 Baseline | 72.21 (8.90) | 72.31 (9.97)
  Week 13 Change from Baseline | 2.05 (10.60) | -0.90 (10.67)
  Week 54 Baseline (n=76, n=90) | 74.95 (10.16) | 71.03 (7.56)
  Week 54 Change from Baseline | -2.46 (10.52) | 1.46 (7.47)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.028, ANOVA — P-value for Week 13 Change from Baseline

18. Secondary Outcome: Change From Baseline to Week 13 and Week 54 Endpoints in Vital Signs: Blood Pressure
Time Frame: Baseline, Week 13, Week 54
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 109 | 116
mm Hg
  Systolic Blood Pressure (SBP) Week 13 Baseline | 127.44 (14.40) | 127.62 (14.75)
  SBP Week 13 Change from Baseline | -0.94 (11.12) | -1.24 (13.30)
  SBP Week 54 Baseline (n=76, n=90) | 127.04 (14.10) | 127.07 (14.99)
  SBP Week 54 Change from Baseline | -1.42 (14.40) | 0.77 (12.98)
  Diastolic Blood Pressure (DBP) Week 13 Baseline | 79.92 (8.63) | 80.38 (8.36)
  DBP Week 13 Change from Baseline | 0.32 (8.27) | -1.25 (7.47)
  DBP Week 54 Baseline (n=76, n=90) | 81.53 (8.19) | 79.74 (8.74)
  DBP Week 54 Change from Baseline | -2.00 (9.37) | 0.50 (8.02)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.764, ANOVA — P-value for SBP Week 13 Change from Baseline
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.093, ANOVA — P-value for DBP Week 13 Change from Baseline

19. Secondary Outcome: Change From Baseline to Week 13 and Week 54 Endpoints in Vital Signs: Weight
Time Frame: Baseline, Week 13, Week 54
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 109 | 116
kilograms (kg)
  Week 13 Baseline | 76.63 (14.83) | 76.29 (14.01)
  Week 13 Change from Baseline | -0.64 (2.32) | 0.08 (1.97)
  Week 54 Baseline (n=81, n=97) | 76.57 (14.61) | 75.34 (13.42)
  Week 54 Change from Baseline | 1.42 (3.25) | -0.38 (2.46)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.008, ANOVA — P-value for Week 13 Change from Baseline

20. Other Pre Specified Outcome: Serious Adverse Events During the Dose-Blind Extension Phase
Description: Serious adverse events during the extension phase reported based on the original treatment group to which the patient was randomized. Dictionary used was MedDRA 11.0.
Time Frame: Week 13 though Week 54
Population: Number of randomized participants who entered the extension phase. Note: Week 54 was the end of the extension phase and all patients received duloxetine - data are reported for all patients who entered extension phase regardless of their original randomization group.
Measure: Number; unit: participants
Arm/Group | Duloxetine
Number analyzed (Participants) | 181
participants
  Patients with ≥1 Serious Adverse Event | 9
  Accidental overdose | 1
  Acute tonsillitis | 1
  Angiopathy | 1
  Back pain | 1
  Femur fracture | 1
  Hand fracture | 1
  Osteoarthritis | 1
  Road traffic accident | 1
  Suicidal ideation | 1
  Syncope | 1
  Tonsillitis | 1

21. Other Pre Specified Outcome: Treatment-Emergent Adverse Events Occurring in at Least 5 Percent of Patients During the Dose-Blind Extension Phase
Description: Treatment-emergent adverse events during the extension phase reported based on the original treatment group to which the patient was randomized. Dictionary used was MedDRA 11.0.
Time Frame: Week 13 through Week 54
Population: as for outcome 20
Measure: Number; unit: participant
Arm/Group | Duloxetine
Number analyzed (Participants) | 181
participant
  Headache | 22
  Nausea | 17
  Abdominal pain upper | 13
  Hyperhidrosis | 11

ADVERSE EVENTS:
Time Frame: Adverse event data in this module is for the 13 Week acute double-blind treatment phase.
Arm/Group | Duloxetine | Placebo
Serious Adverse Events (participants affected / at risk) | 5/115 | 1/121
Other Adverse Events (participants affected / at risk) | 72/115 | 59/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine (N=115) | Placebo (N=121)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Hypertensive encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine (N=115) | Placebo (N=121)
Tachycardia (Cardiac disorders) | 3 (3) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 3 (3) | 0 (0)
Thyroid disorder (Endocrine disorders) | 0 (0) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (3) | 2 (2)
Constipation (Gastrointestinal disorders) | 6 (6) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 8 (9) | 6 (7)
Dry mouth (Gastrointestinal disorders) | 11 (11) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 14 (14) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)
Asthenia (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 8 (9) | 1 (1)
Influenza (Infections and infestations) | 4 (4) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (3) | 3 (4)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2)
Weight increased (Investigations) | 2 (2) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Dizziness (Nervous system disorders) | 7 (7) | 2 (2)
Dysgeusia (Nervous system disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 4 (6) | 12 (14)
Migraine (Nervous system disorders) | 3 (3) | 1 (1)
Somnolence (Nervous system disorders) | 6 (6) | 1 (1)
Insomnia (Psychiatric disorders) | 5 (5) | 5 (5)
Erectile dysfunction (Reproductive system and breast disorders) | 3 (3) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 8 (9) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days